CLINICAL TRIAL: NCT06147258
Title: The Impact of Expressive Emotional Writing on Facilitating Grief Resolution in Adults With Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency)
Responsible Party: Principal Investigator, Hon K. Yuen, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1925594-38; 1925594-38 (Other Grant/Funding Number: National Endowment for the Arts)
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Transverse Myelitis
MeSH Terms: conditions — Spinal Cord Injuries; Myelitis, Transverse

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors are masked to participant group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive writing (Experimental): Participation in a 10 weekly virtual expressive writing with 1 session per week
  Interventions: Behavioral: expressive writing
- Waitlist control (No Intervention): Participation in usual daily activities

INTERVENTIONS:
Behavioral: expressive writing — A typical session will begin with the teaching artist (i.e., writing coach) introducing a new writing theme. Participants will have at least 20 minutes to write, and each session will include post-writing reflections and sharing, an undirected supportive interaction among participants.
  Arms: Expressive writing

SUMMARY:
The aim of this study is to evaluate the therapeutic benefits of a 10-week online coach-guided EEWP on psychosocial health among adults with SCI.

DETAILED DESCRIPTION:
Paralysis in people with spinal cord injury (SCI) leads to grief from the loss of physical capacity, social or occupational role function, and life goals. Expressive emotional writing (EEW) provides an outlet for these individuals to explore and express feelings and emotions that arise from their losses related to limb paralysis. Using a randomized controlled trial design, the proposed project will attempt to confirm the benefits of an online coach-guided EEW program for improving psychosocial health among adults with SCI. Benefits of participating in the program will be evaluated using validated assessments to measure reduction of grief intensity and improvement in other psychosocial dimensions and social participation.

ELIGIBILITY:
Inclusion Criteria: (1) diagnosis (with evidence) of SCI (traumatic or non-traumatic) with limb weakness; (2) aged > 18 years; (3) access to the internet and a computer or to a smartphone that can perform videoconferencing, (4) sufficient English language and cognitive proficiency to complete self-report study questionnaires and understand program content in English, and able to communicate verbally or through writing.

-

Exclusion Criteria: (1) severe cognitive impairments that prevent online learning and completion of the evaluation; (2) suicidal intent requiring emergency care; (3) consistent psychotherapy within the last 6 months; (4) current or planned participation in psychological therapy or a clinical trial during the study period that could affect the outcomes of the study; or (5) congenital SCI (e.g., spinal bifida)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Grief and Loss Scale | baseline, 11 weeks, 3-month follow-up
  a 9-item measure of an individual's emotional reactions or grief such as anger, guilt, anxiety, sadness, and despair in the past 7 days, using a 5-point scale: 1=never to 5=always. The scores range from 9 to 45. Higher scores reflect higher degree of grief and loss.
Impact of Events Scale | baseline, 11 weeks, 3-month follow-up
  a 6-item measure of an individual's distress related to different difficulties in the past 7 days, using a 5-point scale: 0=not at all to 4=extremely. The scores range from 0 to 24. Higher scores reflect greater distress.
Emotional Distress - Depression | baseline, 11 weeks, 3-month follow-up
  It is a part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It is an 8-item measure of an individual's emotional distress (depression) in the past 7 days, using a 5-point scale: 1=never to 5=always. The scores range from 8 to 40. Higher scores reflect higher degree of emotional distress (depression)
Perceived Stress Scale (PSS) | baseline, 11 weeks, 3-month follow-up
  is a 10-item measure of frequency of an individual experiencing stress in the past month, using a 5-point scale: 1=never to 5=very often. Four positively stated items require reversed coding. The scores range from 10 to 50. Higher scores reflect higher frequency of experiencing stress.
Sleep Disturbance | baseline, 11 weeks, 3-month follow-up
  It is a part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It is a 4-item measure of an individual's sleep problem or quality in the past 7 days, using a 5-point scale: 1=not at all to 5=very much or 1=very good to 5=very poor. Two positively stated item require reversed coding. The scores range from 4 to 20. Higher scores reflect greater sleep problem.
Sleep Impact | baseline, 11 weeks, 3-month follow-up
  It is a part of the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ). It is a 5-item measure of an individual's trouble falling asleep in the past 7 days, using a 5-point scale: 5=never to 5=always. One positively stated item require reversed coding. The scores range from 5 to 25. Higher scores reflect less trouble falling asleep.
Meaning and Purpose | baseline, 11 weeks, 3-month follow-up
  It is part of the NIH Toolbox Item Bank. It is a 7-item measure of an individual's meaning and purpose in life, using a 5-point scale:1=strongly disagree to 5=strongly agree. The scores range from 7 to 35. Higher scores reflect greater meaning and purpose in life.
Self-Efficacy for Managing Chronic Conditions - Managing Emotions | baseline, 11 weeks, 3-month follow-up
  It is a part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It is a 4-item measure of an individual's self-efficacy for managing chronic conditions, using a 5-point scale: 1=I am not at all confident to 5=I am very confident. The scores range from 4 to 20. Higher scores reflect greater confident in managing chronic conditions.
Ability to Participate in Social Roles and Activities | baseline, 11 weeks, 3-month follow-up
  It is a 4-item measure of an individual's trouble participating in social roles and activities, using a 5-point scale:1=always to 5=never. The scores range from 4 to 20. Higher scores reflect less trouble participating in social roles and activities.
Satisfaction with Social Roles and Activities | baseline, 11 weeks, 3-month follow-up
  It is a 4-item measure of an individual's satisfaction with social roles and activities, using a 5-point scale:1=not at all to 5=very much. The scores range from 4 to 20. Higher scores reflect greater satisfaction with social roles and activities.
Connor-Davidson Resilience Scale | baseline, 11 weeks, 3-month follow-up
  It consists of 10 statements that respondents rated on a 5-point scale from 0 - Not true at all.
  1 - Rarely true.2 - Sometimes true.3 - Often true.4 - True nearly all the time. Answers were scored from 0 to 4 to create a total score that ranged from 0 to 100, with higher numbers denoting greater resilience.
Cortisol level | baseline, 11 weeks, 3-month follow-up
  Hair cortisol level

CONTACTS AND LOCATIONS:
Overall Officials: Hon Yuen, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States